CLINICAL TRIAL: NCT06473701
Title: BONG: Reducing Severe Breathlessness With Dronabinol in the Severe and Very Severe Chronic Obstructive Pulmonary Disease Patient Group - A Randomized, Double-Blind, Placebo-Controlled, Crossover Study
Brief Title: Reducing Breathlessness With Dronabinol in COPD Patients
Acronym: BONG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); University of Southern Denmark (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2024-513593-22-00
Record Dates: First submitted 2024-05-22; First posted 2024-06-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: COPD; Breathlessness; Cannabis
Keywords: Randomized, Controlled, Double-blind, Crossover trial; Cannabis-based medicine; Cannabis; COPD; Breathlessness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, double-blind, crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An external party will manage the randomization process, assigning participants equally to either the active treatment or placebo groups in a 1:1 ratio. The randomization will be conducted using www.sealedenvelope.com and will incorporate varying block sizes, such as 4, 6, and 8 participants per block. Consequently, each medication container will be labeled with a unique participant number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol 20 mg, then placebo (Experimental): In this arm, the study subject will first receive dronabinol 2.5 mg capsules. For two weeks the subject will titrate dose with one capsule corresponding to 2.5 mg dronabinol every other day until 20 mg. Doses are divided into three times a day. After up titration the subject will receive 20 mg daily treatment over a period of 2 weeks. After a wash out period of 2 weeks, study subject will receive placebo capsules (matching dronabinol 2.5 mg capsules). For two weeks the subject will titrate with one capsule every other day until 20 mg. Doses are divided into three times a day. After up titration the subject will receive 8 daily placebo capsules over a period of 2 weeks.
  Interventions: Drug: Dronabinol 2.5mg Capsule; Drug: Placebo
- Placebo, then dronabinol 20 mg (Placebo Comparator): In this arm, the study subject will first receive placebo capsules (matching dronabinol 2.5 mg capsules). For two weeks the subject will titrate with one capsule every other day until 20 mg. Doses are divided into three times a day. After up titration the subject will receive 8 daily placebo capsules over a period of 2 weeks. After a wash out period of 2 weeks, study subject will receive dronabinol 2.5 mg capsules. For two weeks the subject will titrate dose with one capsule corresponding to 2.5 mg dronabinol every other day until 20 mg. Doses are divided into three times a day. After up titration the subject will receive 20 mg daily treatment over a period of 2 weeks.
  Interventions: Drug: Dronabinol 2.5mg Capsule; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 2.5mg Capsule — Dronabinol 2.5 mg pr capsule. Titration up till 20 mg daily dose.
  Other Names: Delta9-tetrahydrocannabinol
Drug: Placebo — Dronabinol-matched placebo capsule containing no active substance.

SUMMARY:
This clinical trial examines whether Dronabinol, which contains the synthetic psychoactive compound tetrahydrocannabinol (THC), can alleviate severe breathlessness in patients with severe and very severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This study is a randomized, controlled, double-blind, crossover trial evaluating the effectiveness of the pharmaceutical drug Dronabinol in patients with severe and very severe COPD.

The researchers will compare the effects of Dronabinol with a placebo (an identical-looking substance that contains no active drug) to determine if Dronabinol reduces breathlessness in COPD patients.

After enrollment, study subjects will undergo four weeks of treatment with both Dronabinol and the placebo in a blinded and randomized sequence. There is a two-week washout period between treatments. During these treatment phases, subjects will complete questionnaires about their daily experiences of breathlessness and wear a watch that records various health parameters.

The study includes eight visits: the initial enrollment and follow-up checks every two weeks. At these visits, subjects undergo tests for lung function and walking distance, and complete health status questionnaires. Additionally, blood samples for THC levels and hair samples for cortisol analysis are collected.

ELIGIBILITY:
Inclusion Criteria:

* Refractory dyspnea despite optimal treatment
* COPD (GOLD 3,4)
* Breathlessness corresponding to mMRC score ≥ 3
* Informed written consent
* Age ≥ 18 years
* Cognitive relevant, of legal age
* Understands and speaks Danish
* For fertile women defined by amenorrhea for less than 12 months: negative HCG before entry into the trial
* For fertile and sexually active subjects: use of safe contraception during medication intake and 4 weeks after: intrauterine device (IUD) or hormonal contraception (oral contraceptive pill, implant, transdermal patch, vaginal ring or depot injection).

Exclusion Criteria:

* Ongoing infection or exacerbation of COPD within the last month (30 days)
* Regular treatment with THC or CBD within 1 month (30 days)
* Life expectancy less than 3 months (90 days)
* Treatment with medicines that, according to the summary of product characteristics, are strong inhibitors or inducers of CYP3A4, CYP2C9 or CYP2C19
* History of or current evidence of significant medical or psychiatric disorder that is considered by the investigator to put the subject at greater risk of experiencing an adverse event
* Current or past substance abuse where the investigator finds it too risky for the subject to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in Numeric Rating Scale score of discomfort of daily breathlessness between active treatment and placebo | Assessed daily in the baseline period and through both treatment periods. Up to 70 days
  Numeric rating scale score range 0-10. Higher score reflects higher discomfort of breathlessness
Difference in Numeric Rating Scale score of breathlessness interference of daily activities between active treatment and placebo | Assessed daily in the baseline period and through both treatment periods. Up to 70 days
  Numeric rating scale score range 0-10. Higher score reflects more breathlessness interference on daily activities
Correlation between breathlessness rated on a daily numeric rating scale in relation to amount of THC blood level of the active treatment period | Assessed daily in the baseline period and through both treatment periods. Up to 70 days
  Numeric rating scale score range 0-10. Higher score reflects higher discomfort of breathlessness
Correlation between breathlessness interference of daily activities rated on a numeric rating scale in relation to amount of THC blood level of the active treatment period | Assessed daily in the baseline period and through both treatment periods. Up to 70 days
  Numeric rating scale score range 0-10. Higher score reflects more breathlessness interference on daily activities

SECONDARY OUTCOMES:
Difference in Multidimensional Dyspnea Profile questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Assesses different dimensions of COPD.
Difference in COPD Assessment Test questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Assesses the severity of physical COPD symptoms.
Difference in Chronic Respiratory Disease Questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  A HRQL tool which incorporates patient perceptions of both physical and emotional health.
Difference in Hospital Anxiety and Depression Scale questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Assess anxiety and depression symptoms in medical patients.
Difference in Medical Research Council Dyspnea Scale questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  A simple and valid method of categorizing patients with COPD in terms of their disability that could be used to complement FEV1 in the classification of COPD severity.
Difference in Epworth Sleepiness Scale questionnaire score between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Assesses person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Difference in the spirometry parameter forced expiratory volume in 1. second (FEV1) between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  The FEV1 indicates the lung tissue's ability to release air during the first second of exhalation.
Difference in the spirometry parameter forced vital capacity (FVC) between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  The FVC indicates the lung tissue's ability to release air during the entire exhalation.
Difference in the spirometry parameter FEV1/FVC (ratio), between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Can indicate an obstructive pattern in the exhalation which are used in the diagnosis of COPD.
Difference in six-minute walk test(6MWT) between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  6 minutes walking test measures breathlessness and performance ability.
Difference Borg dyspnea score conducted in relation to 6MWT between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  A numeric scale from 0 (no breathlessness) to 10 (extremely strong breathlessness) but not limited to 10 if subjects feel breathlessness above 10
Difference in cortisol level in the hair samples between active treatment and placebo period | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  Measurement of stress through cortisol levels in the hair.

OTHER OUTCOMES:
Difference in clinical parameters between active treatment and placebo period using a yet unspecified continuous monitoring device. | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  For several days in each treatment period we continuously measure blood oxygen saturation, electrodermal activity, pulse rate, sleep recording, temperature, respiratory rate, and activity counter.
Difference in stand-to-sit-test between active treatment and placebo | Baseline (T1; day 1) and after each treatment period (T4; day 28, T7; day 70)
  A measurement for physical capability until breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hilberg, Prof., MD, Principal Investigator — Medical Department, Vejle Hospital
Locations (1):
- Vejle Hospital - A part of Lillebaelt Hospital, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No
It is the plan to share SAP when this is finalized. It is undecided whether CSR and analytic code will be shared on a platform or available on reasonable request.